CLINICAL TRIAL: NCT07008092
Title: Prostaglandin-E Urinary Metabolite (PGE-M) as a Predictor of Acute Appendicitis in Children
Status: Recruiting | Type: Observational
Sponsor: KBC Split (Other)
Responsible Party: Principal Investigator, Tomislav Žuvela, Doctor of Medicine, Plastic surgery resident, KBC Split
Other Study IDs: 2181-147/01-06/LJ.Z.-25-02
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Acute Appendicitis; Acute Appendicitis With Rupture; Abdominal Pain (AP)
Keywords: Acute appendicitis; PGE-M; Prostaglandin-E urinary metabolite
MeSH Terms: conditions — Appendicitis; Abdominal Pain | interventions — Blood Specimen Collection; Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Acute appendicitis with rupture
  Interventions: Diagnostic Test: Blood specimen collection; Diagnostic Test: Urine collection
- Acute appendicitis without rupture
  Interventions: Diagnostic Test: Blood specimen collection; Diagnostic Test: Urine collection
- Control group: Patients with abdominal pain in which acute appendicitis has been ruled out as a cause
  Interventions: Diagnostic Test: Blood specimen collection; Diagnostic Test: Urine collection

INTERVENTIONS:
Diagnostic Test: Blood specimen collection — Blood specimen collection for analysis of C-reactive protein, white blood cell count and neutrophile count.
Diagnostic Test: Urine collection — Urine sample collection for analysis of creatinine and prostaglandin E urinary metabolites

SUMMARY:
Diagnosing acute appendicitis in children remains a clinical challenge, with delayed or incorrect diagnosis potentially leading to serious complications or unnecessary surgery. Prostaglandin E urinary metabolites (PGE-M) have been found elevated in various inflammatory conditions, but their diagnostic value in pediatric appendicitis is not well established. This study aims to assess the potential of PGE-M as a biomarker for acute appendicitis in children.

The study will be conducted over 12 months and will include 100 children aged 5 to 17 years presenting with acute abdominal pain. In addition to routine laboratory tests, urinary PGE-M levels will be analyzed. The study involves minimal risk to participants

DETAILED DESCRIPTION:
The diagnosis of acute appendicitis in children remains a challenge, even for experienced clinicians. Failure to recognize this acute condition may result in perforation and subsequent peritonitis, whereas misdiagnosis can lead to unnecessary (negative) appendectomies. Elevated levels of prostaglandin E urinary metabolites (PGE-M) have been observed in other inflammatory conditions such as inflammatory bowel disease, acute mesenteric ischemia, and necrotizing enterocolitis.

The aim of this study is to determine whether PGE-M levels are elevated in children with acute appendicitis and whether this biomarker could be used in the diagnosis of acute appendicitis.

The planned duration of the study is 12 months, with a projected sample size of 100 participants.

Inclusion criteria: Children aged 5 to 17 years presenting with acute abdominal pain and signs and symptoms suggestive of acute appendicitis, without significant comorbidities.

Exclusion criteria: Children outside the specified age range, those with a previously diagnosed chronic or malignant disease, a history of abdominal surgery, or pregnancy.

For each child included in the study, demographic data, clinical characteristics, laboratory and diagnostic test results, intraoperative findings, and discharge diagnoses will be recorded. Since the child is already indicated for surgery or hospital admission regardless of study participation, there are no significant risks associated with participation in this study-apart from potential, but rare, complications related to peripheral venous blood sampling (e.g., hematoma or discomfort).

For the purposes of the study, a peripheral venous blood sample will be collected (on the day of surgery or hospital admission) to analyze laboratory parameters including leukocyte count, C-reactive protein, and neutrophils. Additionally, a urine sample will be collected to determine the levels of prostaglandin E urinary metabolites (PGE-M) and creatinine

ELIGIBILITY:
Inclusion Criteria:

* children of age 5 -17 years with acute abdominal pain
* children with clinical signs of acute appendicitis

Exclusion Criteria:

* previous diagnosis of chronic and/or malignant disease
* children who had previous abdominal surgery
* pregnancy

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients from 5 to 17 years of age, presenting with acute abdominal pain consistent with diagnosis of acute appendicitis, to Emergency Surgical Department at the University Hospital of Split
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-02 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
PGE-M | 72 hours
  Levels of prostaglandin E urinary metabolite as measured with ELISA test

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Split, Split, Croatia

IPD SHARING:
Plan to Share IPD: No